CLINICAL TRIAL: NCT04664231
Title: The Investigation of the Scoliosis of Children With Juvenile Idiopathic Arthritis and Awareness of the Parents Related to Scoliosis
Brief Title: Spine Deformities in Juvenile Idiopathic Arthritis
Acronym: Scoliosis
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eylül Pınar KISA, Lecturer, Biruni University
Other Study IDs: Pre-PHD thesis
Record Dates: First submitted 2020-11-29; First posted 2020-12-11 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Scoliosis; Juvenile Idiopathic Arthritis; Awareness
Keywords: scoliosis; Juvenile idiopathic arthritis; Awareness; spine
MeSH Terms: conditions — Scoliosis; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with JIA: Children with JIA coming to clinic
- Healthy Children: Healthy Children in the school

SUMMARY:
Juvenile Idiopathic Arthritis (JIA)is the most common chronic rheumatic disease in childhood. While JIA usually affects the ankle and knee joints, it can also affect hip, cervical spine and shoulder involvement. Secondary problems such as spine involvement or lack of weight transfer may lead to scoliosis. The aim of this study was to perform scoliosis screening in children with JIA and to evaluate families' awareness of scoliosis.

DETAILED DESCRIPTION:
Juvenile Idiopathic Arthritis (JIA)is the most common chronic rheumatic disease in childhood. While JIA usually affects the ankle and knee joints, it can also affect hip, cervical spine and shoulder involvement. Secondary problems such as spine involvement or lack of weight transfer may lead to scoliosis. The aim of this study was to perform scoliosis screening in children with JIA and to evaluate families' awareness of scoliosis. aged 4-16 years will include in the study. Trunk rotation measure with scoliometer by applying forward bending test. Children with more than 5 rotations will send to the X-ray. 28 questions will asked, which evaluate the demographic characteristics of children, their educational status, their participation in sports activities, and the physical appearance of families about their children. These questions will asked if the parents had heard of scoliosis before, where they heard it, and whether anyone had scoliosis in the family. Families who complained of posture disorder will asked which shoulder is high without looking at their children and whether they see any height when they leaned forward and the pain situation in their children. Statistical analysis of the data using the SPSS 24.0 (Statistical Package for Social Sciences) program. In all analyzes, p≤0.05 consider statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with rheumatology age between 6-16,
* to be diagnosed at least 6 months ago;
* ability to walk independently; ability to read and write in Turkish; able to follow simple instructions
* no pathology in visual ability and hearing

Exclusion Criteria:

* a history of specific balance problems (i.e., diagnosed vestibular or neurological disorder);
* severe musculoskeletal, neurological or cardiovascular disorders that limit mobility;
* use of medication(s) such as sedatives and hypnotics, antidepressants and benzodiazepines
* participate in scoliosis rehabilitation in the lasts 6-months.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with juvenile idiopathic arthritis
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Assesment of angle of trunk rotation | Baseline
  Angle of trunk rotation (ATR) will be evaluated with Scoliometer.It is an easy-to-use, reliable, practical specially designed inclinometer for scoliometer. The evaluation will be done with Adam's Bend test, in the standing forward bending position. Child's feet will be positioned parallel to each other. The physiotherapist who measures to adjust the distance between the feet, by placing one foot between the two feet of the child, by moving the scoliometer from the beginning of the thoracic to the sacrum, the largest measured angle of rotation will be recorded.
Radiological imaging | Baseline
  Radiological imaging shows vertebrae' lateral tilt degree. It calculated with Cobb angle method. The Cobb angle provides information about the degree of scoliosis.i It is accepted as a clinical evaluation method used in giving information about scoliosis and determining the effectiveness of treatment and prognosis of scoliosis.

SECONDARY OUTCOMES:
Patient awareness forms | Baseline
  It will be created to obtain sociodemographic information and personal data about the disease. In this context, gender, age, height, weight, occupation, educational status, dominant side, affected side (s) and patient history, disease duration, time spend at the desk and sports activity will be questioned in detail. For family Scoliosis Awareness, Have you heard of scoliosis?, Is there a family?, Are the child's shoulder heights equal? (Say without looking), Which one is high? When you bend forward, do you see an asymmetry on the back?, Is there any pain? questions will ask

CONTACTS AND LOCATIONS:
Overall Officials: KISA, Study Director — Biruni University
Locations (1):
- Eylül Pınar Kısa, Istanbul, Turkey (Türkiye)